CLINICAL TRIAL: NCT05240976
Title: Combination of NMDA-enhancing and Anti-inflammatory Treatments for Ultra-resistant Schizophrenia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMUH109-REC3-043
Record Dates: First submitted 2022-01-24; First posted 2022-02-15 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Schizophrenia
Keywords: Ultra-resistant schizophrenia; NMDA; Inflammation
MeSH Terms: conditions — Schizophrenia; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMDAE plus Anti-inflammatory Agent (AIFA) (Experimental): An NMDA enhancer plus a drug with anti-inflammatory property
  Interventions: Drug: NMDAE plus AIFA
- NMDAE plus Placebo (Placebo Comparator): An NMDA enhancer plus Placebo
  Interventions: Drug: NMDAE plus Placebo Cap

INTERVENTIONS:
Drug: NMDAE plus AIFA — Use of an NMDA enhancer plus a drug with anti-inflammatory property for the treatment of ultra-resistant schizophrenia.
  Arms: NMDAE plus Anti-inflammatory Agent (AIFA)
Drug: NMDAE plus Placebo Cap — Use of an NMDA enhancer plus placebo as a comparator
  Arms: NMDAE plus Placebo

SUMMARY:
Previous study found that some NMDA-enhancing agent was able to augment efficacy of clozapine for clinical symptoms but not cognitive function in the treatment of ultra-resistant schizophrenia. In addition, several drugs with anti-inflammatory properties have been tested in clinical trials for the treatment of schizophrenia. Whether a drug with anti-inflammatory property can strengthen the efficacy of an NMDA-enhancer (NMDAE) in the treatment of ultra-resistant schizophrenia remains unknown.

DETAILED DESCRIPTION:
Several lines of evidence suggest that both NMDA and inflammatory hypotheses have been implicated in schizophrenia. Previous study found that some NMDA-enhancing agent was able to augment efficacy of clozapine for clinical symptoms but not cognitive function in the treatment of ultra-resistant schizophrenia. In addition, several drugs with anti-inflammatory properties have been tested in clinical trials for the treatment of schizophrenia. Whether a drug with anti-inflammatory property can strengthen the efficacy of an NMDA-enhancer (NMDAE) in the treatment of ultra-resistant schizophrenia remains unknown.

Therefore, this study aims to compare NMDAE plus a drug with anti-inflammatory property and NMDAE plus placebo in the treatment of ultra-resistant schizophrenia. The subjects are the patients with ultra-resistant schizophrenia who have responded poorly to clozapine treatment. They keep their original clozapine treatment and are randomly, double-blindly assigned into two treatment groups for 12 weeks: (1) NMDAE plus Anti-inflammatory Agent (AIFA), or (2) NMDAE plus placebo. Cognitive functions are assessed at baseline and at endpoint of treatment by a battery of tests. Clinical performances and side effects are measured at weeks 0, 2, 4, 6, 9, and 12. The efficacies of NMDAE plus AIFA and NMDAE plus placebo will be compared.

Chi-square (or Fisher's exact test) will be used to compare differences of categorical variables and t-test (or Mann-Whitney test if the distribution is not normal) for continuous variables between treatment groups. Mean changes from baseline in repeated-measure assessments will be assessed using the generalized estimating equation (GEE) for both primary and secondary outcomes . All p values for clinical measures will be based on two-tailed tests with a significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Have a DSM-5 (American Psychiatric Association) diagnosis of schizophrenia
* Are treatment-resistant to standard treatments of at least two specific antipsychotics before clozapine treatment
* Are receiving adequate trials of clozapine for more than 12 weeks but without satisfactory response
* PANSS total score ≥ 70; SANS total score ≥ 40
* Have sufficient education to communicate effectively and are capable of completing the assessments of the study
* Agree to participate in the study and provide informed consent

Exclusion Criteria:

* DSM-5 diagnosis of intellectual disability or substance (including alcohol) use disorder
* History of epilepsy, head trauma, or serious medical or central nervous system diseases (other than schizophrenia) which may interfere with the study
* Clinically significant laboratory screening tests (including blood routine, biochemical tests)
* Pregnancy or lactation
* Inability to follow protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change of cognitive function | Week 0, 12
  The measure is the composite from multiple measures. All tests have no unit. For the domain (a. and c.) with more than one test, a composite T score will be calculated by standardizing the average of each T score. Furthermore, a global composite score (for all seven domains) and a neurocognitive composite score (for the first 6 domains) will be also calculated by standardizing the average of the T score of each domain (Lane HY et al, JAMA Psychiatry 2013).
  Ten tests for assessing 7 cognitive domains:
  1. speed of processing (assessed by Category Fluency, Trail Marking A, WAIS-III Digit Symbol-Coding);
  2. sustained attention (Continuous Performance Test);
  3. working memory: verbal (digit span) and nonverbal (spatial span);
  4. verbal learning and memory (WMS-III, word listing);
  5. visual learning and memory (WMS-III, visual reproduction);
  6. reasoning and problem solving (WISC-III, Maze);
  7. social cognition (MSCEIT Version 2)

SECONDARY OUTCOMES:
Change of Positive and Negative Syndrome Scale (PANSS) | week 0, 2, 4, 6, 9, 12
  Assessment of overall symptoms. Minimum value: 30, maximum value:210, the higher scores mean a worse outcome.
  As shown in "Detailed Description", "mean changes from baseline in repeated-measure assessments will be assessed using the generalized estimating equation (GEE) for both primary and secondary outcomes. That is, GEE is used for analyzing the changes from baseline in repeated-measure assessments by a single analysis (but not multiple analyses).
Change of scale for the Assessment of Negative Symptoms (SANS) total score | week 0, 2, 4, 6, 9, 12
  Assessment of negative symptoms. Minimum value: 0, maximum value:100, the higher scores mean a worse outcome.
Chang of positive subscale of PANSS | week 0, 2, 4, 6, 9, 12
  Assessment of positive symptoms. Minimum value: 7, maximum value:49, the higher scores mean a worse outcome.
Change of negative subscale of PANSS | week 0, 2, 4, 6, 9, 12
  Assessment of negative symptoms. Minimum value: 7, maximum value:49, the higher scores mean a worse outcome.
Change of general Psychopathology subscale of PANSS | week 0, 2, 4, 6, 9, 12
  Assessment of general psychopathology. Minimum value: 16, maximum value:112, the higher scores mean a worse outcome
Change of clinical Global Impression | week 0, 2, 4, 6, 9, 12
  Assessment of general impression. Minimum value: 1, maximum value:7, the higher scores mean a worse outcome.
Change of global Assessment of Functioning | week 0, 2, 4, 6, 9, 12
  Assessment of social, occupational, and psychological function. Minimum value: 1, maximum value:100, the higher scores mean better function.
Change of hamilton Rating Scale for Depression | week 0, 2, 4, 6, 9, 12
  Assessment of depressive symptoms. Minimum value: 0, maximum value:52, the higher scores mean a worse outcome.
Change of quality of Life Scale | week 0, 2, 4, 6, 9, 12
  Assessment of life quality. Minimum value: 0, maximum value:126, the higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, China Medical University Hospital, Taichung, Taiwan